CLINICAL TRIAL: NCT07406815
Title: The Value of Near-Infrared Fluorescence Imaging in the Protection of the Recurrent Laryngeal Nerve During Minimally Invasive Esophagectomy：A Prospective Randomized Controlled Trial
Brief Title: The Value of Near-Infrared Fluorescence Imaging in the Protection of the Recurrent Laryngeal Nerve During Minimally Invasive Esophagectomy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NERV-ICG
Record Dates: First submitted 2024-11-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer; Recurrent Laryngeal Nerve; ICG (Indocyanine Green); Lymph Node Dissection
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (ICG group) receiving VATS with near-infrared-indocyanine green fluorescence for RLN visualization (Experimental)
  Interventions: Drug: ICG (Indocyanine Green)
- (Control group) receiving VATS without near-infrared-indocyanine green fluorescence for RLN visualiz (No Intervention)

INTERVENTIONS:
Drug: ICG (Indocyanine Green) — Minimally invasive surgery for esophageal cancer using near-infrared indocyanine green fluorescence to visualize the recurrent laryngeal nerve.
  Arms: (ICG group) receiving VATS with near-infrared-indocyanine green fluorescence for RLN visualization

SUMMARY:
The goal of this clinical trial is to learn whether the application of indocyanine green near-infrared imaging system can accurately locate the recurrent laryngeal nerve (RLN) during lymph node dissection in esophageal cancer radical surgery, thereby reducing the risk of RLN injury. The main questions it aims to answer are:

1. Can preoperative intravenous administration of indocyanine green enable visualization of the RLN;
2. Does performing RLN dissection guided by near-infrared imaging system reduce the probability of RLN injury, leading to better clearance of RLN lymph nodes and improved RLN protection rates? Researchers will compare whether indocyanine green was intravenously administered preoperatively to assess intraoperative RLN visualization. Participants in the study group will receive intravenous indocyanine green at a dose of 5mg/kg 24 hours before surgery. All patients will be monitored for RLN injury-related complications postoperatively, and RLN injury status will be objectively assessed via laryngoscopy one week post-operation.

DETAILED DESCRIPTION:
Surgical treatment is currently the best and preferred method for treating esophageal cancer. Esophagectomy is a highly specialized surgery with a high incidence of complications, among which recurrent laryngeal nerve (RLN) paralysis is one of the most common postoperative complications, severely affecting postoperative quality of life. This study adopts a single-center, prospective, open, controlled, non-inferiority validation design. It focuses on patients with esophageal cancer scheduled for esophageal cancer radical surgery. The study aims to include 144 patients with esophageal cancer, randomized in a 1:1 ratio into two groups: the experimental group receiving indocyanine green (ICG) injection and the control group not receiving ICG injection. A comparison will be made between the two groups regarding laryngeal physiological changes one week post-operation. The study will observe the occurrence rate of symptoms related to RLN injury post-surgery, the duration of RLN dissection, and other relevant indicators. The goal is to explore whether the application of NIR-ICG imaging systems can accurately locate the RLN during lymph node dissection in esophageal cancer radical surgery, thereby reducing the risk of RLN injury.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years at the time of diagnosis (excluding 18 and 75);
* Preoperative biopsy pathology confirming esophageal cancer;
* Undergoing elective thoracoscopic esophageal cancer radical surgery with intraoperative anastomosis;
* Tolerable heart, lung, liver, and kidney function for surgery;
* Patients and their families are able to understand and willing to participate in this clinical study, and have signed an informed consent form.

Exclusion Criteria:

* Allergy to ICG or iodine;
* History of neck or thoracic surgery;
* Patients requiring emergency surgery;
* Tumors involving adjacent organs necessitating combined organ resection;
* Patients with tumor recurrence or distant metastasis;
* Participation in or having participated in other clinical trials within 4 weeks prior to selection;
* History of severe mental illness;
* Pregnant or lactating women;
* Patients with other conditions deemed unsuitable for participation by the investigator;
* Intraoperative conversion to open thoracotomy.
* Patients who, after assessment or intraoperative exploration, cannot undergo the planned surgery;
* Patients who voluntarily withdraw from the study;
* Patients with concomitant non-neoplastic conditions that prevent them from continuing with the study protocol;
* Patients who, after enrollment in the study, are unable to complete it due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Recurrent Laryngeal Nerve Injury | From enrollment to the end of surgery at 1 weeks
  Definition and Significance: This is the core indicator for verifying the research hypothesis. It refers to the proportion of patients with objectively confirmed unilateral or bilateral RLN dysfunction after radical esophagectomy for esophageal cancer. The difference in this incidence between the ICG fluorescence-guided group and the conventional surgery (control) group will be compared.
  Assessment Method:Performed 7 days postoperatively (allowing for resolution of acute edema) by an independent otolaryngologist or speech-language pathologist blinded to the patient's group assignment, using fiberoptic laryngoscopy.
  Quantitative Indicators: Incidence=(Number of patients diagnosed with RLN palsy in each group / Total number of patients in that group) × 100%.

SECONDARY OUTCOMES:
Rates of Temporary vs. Permanent RLN Injury | Repeat fiberoptic laryngoscopy at 1, 3, 6, and 12 months postoperatively.
  Definition: Distinguishes the nature of nerve injury. Temporary injury refers to nerve function that recovers within 6 months postoperatively; permanent injury refers to function that has not recovered after 6 months.
  Assessment Method: Repeat fiberoptic laryngoscopy at 1, 3, 6, and 12 months postoperatively.
  Quantitative Indicators: Calculate the proportion of temporary and permanent injuries both among total injuries and among the total patient population.
Incidence and Severity of Postoperative Voice Dysfunction | 1 month after surgery
  Definition: Assesses the functional consequences resulting from RLN injury.
  Assessment Method:
  (1) Voice Assessment: Use validated patient-reported questionnaires, such as the Voice Handicap Index-10 (VHI-10).
  【Tips: The Voice Handicap Index-10 (VHI-10) has a score range of 0 to 40; a higher score indicates that voice handicap has a greater impact on daily life.】
  Quantitative Indicators:
  (1) Proportion of patients with a VHI-10 total score ≥ 15 (indicating moderate or worse voice handicap) at a specified postoperative timepoint (e.g., 1 month).
Number of Lymph Nodes Dissected in the RLN Region | 1 week after surgery.
  Definition: Verifies whether ICG-guided nerve preservation compromises the oncological radicality of lymphadenectomy.
  Assessment Method: Based on the final postoperative pathological report.
  Quantitative Indicators:
  (1) Total Number of lymph nodes harvested from the bilateral RLN regions (left + right) per group.
Incidence of Postoperative Pulmonary Complications | 30 days after surgery.
  Definition: RLN injury predisposes to aspiration and pneumonia, making this a crucial clinical safety indicator.
  Assessment Method: Use standardized definitions, such as the Clavien-Dindo classification or the Esophagectomy Complications Consensus Group (ECCG) definitions, to record pneumonia, respiratory failure, ARDS, etc., occurring within 30 days postoperatively.
  Quantitative Indicators: Proportion of patients experiencing pulmonary complications of Grade II or higher.
Incidence and Severity of Postoperative Swallowing Dysfunction | 30 days after surgery
  Definition: Assesses the functional consequences resulting from RLN injury.
  Assessment Method:
  (1) Swallowing Assessment: Use the M.D. Anderson Dysphagia Inventory (MDADI). 【Tips: MDADI consists of 20 items and covers four domains: global, emotional, functional, and physical. It uses a 5-point Likert scale for scoring, and both the domain scores and the total score range from 0 to 100 points. A higher score indicates better swallowing function and quality of life.】
  Quantitative Indicators:
  (1) Inter-group comparison of MDADI total scores or subscale scores.
Postoperative Hospital Stay Length | 30 days after surgery.
  Definition: Reflects the overall recovery profile after surgery.
  Quantitative Indicators:
  (1) Postoperative Length of Stay (LOS): Number of days from surgery to meeting discharge criteria.
Quality of Lymph Nodes Dissected in the RLN Region | 1 week after surgery.
  Definition: Verifies whether ICG-guided nerve preservation compromises the oncological radicality of lymphadenectomy.
  Assessment Method: Based on the final postoperative pathological report.
  Quantitative Indicators:
  (1) Metastasis Positive Rate in this region (number of metastatic lymph nodes / total number harvested).
Postoperative Readmission Rate. | 30 days after surgery.
  Definition: Reflects the overall recovery profile after surgery.
  Quantitative Indicators:
  (1) 30-day Unplanned Readmission Rate: Particularly the rate of readmission due to pneumonia, dysphagia, or hoarseness-related issues.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Taniyama Y, Miyata G, Kamei T, Nakano T, Abe S, Katsura K, Sakurai T, Teshima J, Hikage M, Ohuchi N. Complications following recurrent laryngeal nerve lymph node dissection in oesophageal cancer surgery. Interact Cardiovasc Thorac Surg. 2015 Jan;20(1):41-6. doi: 10.1093/icvts/ivu336. Epub 2014 Oct 13. PMID 25312996
- [Result] Bundred JR, Hollis AC, Evans R, Hodson J, Whiting JL, Griffiths EA. Impact of postoperative complications on survival after oesophagectomy for oesophageal cancer. BJS Open. 2020 Jun;4(3):405-415. doi: 10.1002/bjs5.50264. Epub 2020 Feb 17. PMID 32064788
- [Result] Gelpke H, Grieder F, Decurtins M, Cadosch D. Recurrent laryngeal nerve monitoring during esophagectomy and mediastinal lymph node dissection. World J Surg. 2010 Oct;34(10):2379-82. doi: 10.1007/s00268-010-0692-0. PMID 20563722
- [Result] Hikage M, Kamei T, Nakano T, Abe S, Katsura K, Taniyama Y, Sakurai T, Teshima J, Ito S, Niizuma N, Okamoto H, Fukutomi T, Yamada M, Maruyama S, Ohuchi N. Impact of routine recurrent laryngeal nerve monitoring in prone esophagectomy with mediastinal lymph node dissection. Surg Endosc. 2017 Jul;31(7):2986-2996. doi: 10.1007/s00464-016-5317-8. Epub 2016 Nov 8. PMID 27826777
- [Result] Chevallay M, Jung M, Chon SH, Takeda FR, Akiyama J, Monig S. Esophageal cancer surgery: review of complications and their management. Ann N Y Acad Sci. 2020 Dec;1482(1):146-162. doi: 10.1111/nyas.14492. Epub 2020 Sep 15. PMID 32935342